CLINICAL TRIAL: NCT00219154
Title: A Twenty Six-week, Randomized, Double-blind, Parallel Group, Multicenter, Active Controlled, Dose Titration Study to Evaluate the Efficacy and Safety of Aliskiren Compared to HCTZ With the Optional Addition of Amlodipine, Followed by a Second Twenty Six Weeks of Blinded Treatment, in Patients With Essential Hypertension
Brief Title: A Clinical Study to Compare Long-term Efficacy and Safety of an Aliskiren Based Regimen to a Hydrochlorothiazidebased Treatment Regimen With Optional Addition of Amlodipine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2323
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
This study is designed to compare the long-term efficacy and safety of an aliskiren based regimen to an HCTZ based treatment regimen with optional addition of amlodipine in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

-Patients with essential hypertension

Exclusion Criteria:

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of myocardial infarction. Other protocol-defined inclusion exclusion criteria also apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1125 (Actual)
Dates: Start 2005-03; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 26 weeks

SECONDARY OUTCOMES:
Change from baseline systolic blood pressure after 26 weeks
Mean sitting diastolic blood pressure < 90 mmHg or a reduction of > 10 mmHg after 26 weeks
Achieve blood pressure of < 140/90 mmHg after 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Schmieder RE, Philipp T, Guerediaga J, Gorostidi M, Smith B, Weissbach N, Maboudian M, Botha J, van Ingen H. Long-term antihypertensive efficacy and safety of the oral direct renin inhibitor aliskiren: a 12-month randomized, double-blind comparator trial with hydrochlorothiazide. Circulation. 2009 Jan 27;119(3):417-25. doi: 10.1161/CIRCULATIONAHA.107.750745. Epub 2009 Jan 12. PMID 19139391